CLINICAL TRIAL: NCT01578291
Title: Parent Education and Medical Play: A Comparison of Psychological Preparation Strategies for Voiding Cystourethrogram
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment was not on target, evised AAP guidelines may have contributed to the decrease in the number of potential participants
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NA_00034999
Record Dates: First submitted 2012-04-10; First posted 2012-04-16 (Estimated); Last update posted 2017-12-11 (Actual); Status verified 2017-12

CONDITIONS: Vesicoureteral Reflux
Keywords: Play therapy; Urinary tract infections; Children; Vesicoureteral reflux
MeSH Terms: conditions — Vesico-Ureteral Reflux; Urinary Tract Infections | interventions — Play Therapy; Behavior Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- No intervention (No Intervention): Parents given routine information by the medical staff.
- Parental information (Active Comparator): Parents are provided with an educational brochure of the study and the expectations of the discomfort.
  Interventions: Behavioral: Parental information; Behavioral: Play therapy
- Play Therapy (Active Comparator): Child and the parents will spend time in the office with the child life therapist undergoing play therapy.
  Interventions: Behavioral: Parental information; Behavioral: Play therapy

INTERVENTIONS:
Behavioral: Parental information — An informational brochure indicating the study details
  Other Names: Informational materials.
  Arms: Parental information; Play Therapy
Behavioral: Play therapy — Play therapy with a child life specialist
  Other Names: Behavioral therapy; Child life intervention
  Arms: Parental information; Play Therapy

SUMMARY:
Hypothesis: The use of parent education and medical play will be able to reduce patient discomfort with potential uncomfortable medical procedures.

Children that have urinary tract infections and those diagnosed with vesicoureteral reflux undergo a procedure called a voiding cystourethrogram (VCUG) to identify and follow vesicoureteral reflux. For many children and parents this can lead to considerable distress. Pre-procedure preparation can potentially reduce anxiety and improve overall experience with the procedure.

DETAILED DESCRIPTION:
Children that are evaluated medically and found to need a VCUG would be eligible for participation in this study. Children would be randomized to having play therapy or a parental education brochure. The study would have no impact on the child recieving the state of the art medical care.

Play therapy involves having the child play through the process of the study with a child life therapist, in an effort to prepare the child for the procedure. Parents/patients will be given a pre and post procedure evaluation form to objectively categorize the parental/patient perception of the experience with the study.

ELIGIBILITY:
Inclusion Criteria:

* Children that have been identified to need a voiding cystourethrogram

Exclusion Criteria:

* Significant medical conditions that preclude child from being able to understand play therapy or have been identified in the past to have so much discomfort from prior studies as to not be able to participate.

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Does Parent Education and Medical play reduce anxiety and discomfort associated with Voiding Cystourethrogam | 12 months anticipated
  Medical play therapy could potentially reduce parental and pateint anxiety when used for preparing children for medical procedures. This study is designed to identify if play therapy can lead to reduction in parental and pateint anxiety with voiding cystourethrogram - a commonly performed test for the evaluation of children with urinary tract infections.

CONTACTS AND LOCATIONS:
Overall Officials: Ranjuv Mathews, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Childrens Center, Baltimore, Maryland, United States